CLINICAL TRIAL: NCT07141784
Title: Combined Virtual Reality-Integrated C-Mill® and Conventional Therapy Improves Walking, Mobility, and Quality of Life After Motor-Incomplete Spinal Cord Injury
Brief Title: VR-Integrated C-Mill® Combined With Conventional Therapy in Motor-Incomplete SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AnkaraCHBilkent-PMR-MSS-04
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Spinal Cord Injury; Gait; C-Mill; Virtual Reality; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C-Mill® Treadmill Training Plus Conventional Physiotherapy (Experimental): Participants received an integrated rehabilitation program consisting of C-Mill® treadmill training combined with conventional physiotherapy. The program lasted 4 weeks and included 10 C-Mill® sessions in addition to individualized physiotherapy exercises. Each C-Mill® session incorporated virtual reality and gamified tasks to improve static and dynamic balance and to regulate gait. Conventional physiotherapy focused on mobility, muscle strength, and functional skills to enhance walking performance and independence.
  Interventions: Device: C-Mill® Treadmill Training Combined with Conventional Physiotherapy

INTERVENTIONS:
Device: C-Mill® Treadmill Training Combined with Conventional Physiotherapy — Participants received a 4-week integrated rehabilitation program consisting of 10 C-Mill® treadmill training sessions in addition to individualized conventional physiotherapy. C-Mill® sessions incorporated virtual reality and gamified tasks to improve static and dynamic balance, gait speed, stride regulation, and safe obstacle negotiation. Conventional physiotherapy targeted mobility, muscle strength, and functional skills to enhance walking performance and independence.

SUMMARY:
This study investigates the effects of C-Mill® treadmill training, which integrates virtual reality and gamified tasks, combined with conventional physiotherapy, on walking ability, mobility, functional independence, and health-related quality of life in individuals with motor-incomplete spinal cord injury (iSCI).

Participants are adults aged 18 years or older with injury at the T4 level or below, classified as American Spinal Injury Association (ASIA) Impairment Scale grade C or D, and with ICD-10 codes S24.73-S24.77 or S34.70. Individuals with a history of osteoporosis, cardiopulmonary disease, other neurological disorders, joint-related conditions, or concurrent participation in another study are excluded.

All participants complete a 4-week integrated rehabilitation program at a specialized spinal cord injury center. The program consists of 10 C-Mill® sessions in addition to conventional physiotherapy, targeting balance, gait, and walking speed through task-specific training and individualized exercises to improve mobility, strength, and functional skills.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) limits mobility and independence, creating substantial physical and psychological burdens. Virtual reality and gamified treadmill systems such as the C-Mill® may enhance walking rehabilitation through task-specific and engaging practice.

This observational study investigated the effects of C-Mill® treadmill training combined with conventional physiotherapy on walking ability, mobility, functional independence, and health-related quality of life in individuals with motor-incomplete SCI (iSCI). The C-Mill® system provides task-specific, engaging, and safe walking practice through real-time visual feedback and interactive scenarios designed to improve balance, gait speed, and obstacle negotiation.

Participants were adults aged 18 years or older, with spinal cord injury at the T4 level or below, classified as American Spinal Injury Association (ASIA) Impairment Scale grade C or D. ICD-10 codes for inclusion ranged from S24.73 to S24.77 or S34.70. Individuals were in the chronic phase of iSCI and were excluded if they had a history of osteoporosis, cardiopulmonary disease, other neurological disorders, joint-related conditions, or concurrent participation in another study.

All participants completed a 4-week integrated rehabilitation program at a specialized spinal cord injury center. The program consisted of 10 C-Mill® training sessions in addition to conventional physiotherapy. Each C-Mill® session included activities targeting static and dynamic balance, stride regulation, and safe gait adaptation, with progressive difficulty tailored to each participant's abilities. Conventional therapy included individualized physiotherapy exercises focusing on mobility, strength, and functional skills to support walking performance and independence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of spinal cord injury at T4 level or lower
* American Spinal Injury Association (ASIA) Impairment Scale classification of grade C or D
* ICD-10 codes S24.73 to S24.77 or S34.70

Exclusion Criteria:

* History of osteoporosis
* Cardiopulmonary disease
* Other neurological disorders
* Joint-related conditions
* Concurrent participation in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 24 months
  Berg Balance Scale for balance assessment

SECONDARY OUTCOMES:
ASIA Lower Extremity Muscle Score | 24 months
  Assessment of lower extremity muscle strength using the American Spinal Injury Association (ASIA) Lower Extremity Motor Score (LEMS)
Timed Up and Go Test | 24 months
  Timed Up and Go Test overground walking assessment
Walking Index in Spinal Cord Injury II | 24 months
  Walking Index in Spinal Cord Injury II for walking independence level assessment
Ten-Meter Walking Test | 24 months
  Ten-Meter Walking Test for overground walking speed assessment
Gait Speed with Treadmill-Based Gait Analysis | 24 months
  Uses treadmill equipment to assess walking speed (kilometers per hour [km/h]) during gait analysis.
Cadence Measurement with Treadmill-Based Gait Analysis | 24 months
  Uses treadmill equipment to assess cadence (number of steps per minute)
Stride Length Measurement with Treadmill-Based Gait Analysis | 24 months
  Uses treadmill equipment to assess the length of a single stride during walking.
Step Width Measurement with Treadmill-Based Gait Analysis | 24 months
  Uses treadmill equipment to assess the distance between the heels of the feet during walking
Stance Time Difference with Treadmill-Based Gait Analysis | 24 months
  Uses treadmill equipment to assess stance time difference between lower limbs (seconds [s]) during gait analysis.
Spinal Cord Independence Measure (SCIM III) | 24 months
  Spinal Cord Independence Measure (SCIM III) for activity of daily living assessment
World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) | 24 months
  World Health Organization Quality of Life Scale-Short Form (WHOQOL - BREF) for quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)